CLINICAL TRIAL: NCT00046709
Title: Marijuana in Combination With Opioids for Cancer Pain: A Pilot Study
Brief Title: Marijuana for Cancer Pain
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued due to non-enrollment.
Sponsor: Center for Medicinal Cannabis Research (Other)
Collaborators: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C00-SF-108; CC#057; NCT00052871 (obsolete NCT alias)
Record Dates: First submitted 2002-10-01; First posted 2002-10-02 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms
Keywords: Cancer pain; All types of cancer except lung cancer
MeSH Terms: conditions — Neoplasms; Cancer Pain

INTERVENTIONS:
Drug: Smoked Marijuana

SUMMARY:
To find out if it is safe and effective to use smoked marijuana in combination with opioids to treat cancer pain. The study will evaluate whether smoked marijuana, when used with opioids, will have an effect on pain relief, and to see if marijuana reduces the side effects of opioids, which include nausea and/or vomiting.

DETAILED DESCRIPTION:
To take part in this study, you must have ongoing cancer pain which is currently being treated with opioids. If you meet all the eligibility criteria you will be admitted to the General Clinical Research Center at San Francisco General Hospital for 9 days. The treatment consists of smoking one marijuana cigarette 3 times a day.

ELIGIBILITY:
INCLUSION CRITERIA

* Have ongoing cancer pain
* Be diagnosed with cancer and have at least a six month survival.
* Be on a stable dose of opioid medication for at least 2 weeks before enrollment.
* Have smoked marijuana on at least 6 occasions in their lifetime prior to enrollment.

EXCLUSION CRITERIA

You must not:

* Start chemotherapy, radiation or biphosphonates during the study, or have received any new intervention with any such agents within the past 4 weeks.
* Currently be using smoked tobacco products.
* Currently be in methadone treatment.
* Have smoked marijuana within 30 days of enrollment.
* Be diagnosed with diabetes mellitus.
* Have severe heart disease, uncontrolled hypertension, or lung disease.
* Currently be receiving treatment with corticosteroids.
* Be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2002-09; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change in level of cancer pain as recorded on a 100mm Visual Analog Scale.

SECONDARY OUTCOMES:
Change in level of experimentally induced pain on a 100mm Visual Analog Scale.
Change in nausea and emesis in participants exhibiting these symptoms.
Change in disposition kinetics of opioid analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, M.D., Principal Investigator — UCSF Community Consortium
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu